CLINICAL TRIAL: NCT05753007
Title: A Randomized, Double-blind, Clinical Trial of a Hemp-Derived, High Cannabidiol Product for Anxiety in Glioblastoma Patients
Brief Title: A Clinical Trial of a Hemp-Derived, High Cannabidiol Product for Anxiety in Glioblastoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by sponsor due to low enrollment.
Sponsor: Mclean Hospital (Other)
Collaborators: University of California, San Francisco (Other); Center for Medicinal Cannabis Research (Other)
Responsible Party: Principal Investigator, Staci Gruber, Ph.D., Director, Marijuana Investigations for Neuroscientific Discovery; Director, Cognitive and Clinical Neuroimaging Core, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-38341
Record Dates: First submitted 2023-02-10; First posted 2023-03-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (CBD) Solution Plus Standard of Care (SOC) (Experimental): Full-spectrum, hemp-derived, ultra-high CBD solution administered for 8 weeks along with standard of care treatment
  Interventions: Drug: Cannabidiol (CBD)
- Placebo (Placebo Comparator): Placebo solution administered for 8 weeks along with standard of care treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Custom-formulated full-spectrum solution high in cannabidiol
  Arms: Cannabidiol (CBD) Solution Plus Standard of Care (SOC)
Drug: Placebo — Placebo solution
  Arms: Placebo

SUMMARY:
Glioblastoma (GBM) is the most common malignant brain tumor among adults. As the diagnosis is generally considered terminal, patients with GBM often suffer from anxiety and other comorbid conditions, including depression, pain, and sleep disturbance, all of which significantly impact their quality of life. Previous studies have demonstrated the potential of cannabinoids, particularly cannabidiol (CBD), to improve the aforementioned symptoms without conferring significant risks or side effects. Further, recent in-vitro and in-vivo work suggests potential cytotoxic and anti-tumor effects of CBD and other cannabinoids.

This study includes a double-blind, placebo-controlled, 8-week randomized clinical trial assessing the impact of a custom formulated, full-spectrum, hemp-derived ultra-high CBD product on measures of anxiety, pain, and quality of life in newly-diagnosed GBM patients undergoing standard of care (SOC) treatment; the impact of this product vs. placebo on tumor progression will also be assessed. The proposed clinical trial will provide important information that does not currently exist regarding the potential efficacy of a novel full-spectrum, ultra-high CBD product to address clinical symptoms in patients with GBM.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of newly diagnosed glioblastoma, evidenced by neuropathology report and based on World Health Organization (WHO) 2021 classification, and who are to undergo SOC (~ 6 weeks of treatment) with radiation and temozolomide (patients using Optune may be included).
* Written informed consent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* Fluent in English.
* Endorses at least moderate levels of anxiety (on the BAI or OASIS) at the screening visit
* Stable medication/psychotherapy regimens for at least 1 month prior to starting the study (excluding new glioblastoma treatment-related medications or radiation).
* Karnofsky Performance Scale (KPS) of 60 or higher.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigators would compromise the safety of the patient or the quality of the data.
* Current substance use disorder, psychotic disorder, bipolar disorder, or eating disorder.
* Current use of recreational cannabis, medical cannabis, or hemp-derived cannabinoid products more frequently than 1x/month; positive urine delta-9 tetrahydrocannabinol (THC) test.
* Presence of a serious or unstable medical illness, including liver, kidney, or cardiovascular disease.
* Current use of valproate (due to potential for drug-drug interactions).
* Currently enrolled in other research studies or clinical trials involving therapeutic interventions.
* Subjects with serum transaminase (ALT, AST, and total bilirubin) levels >3 times upper limit of normal (UNL) <24 hours prior to day 1 of treatment.
* Contraindication to MRI such as non-MR conditional medical devices or ferrous retained foreign bodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-02-11 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-Reported Anxiety as Assessed by the Beck Anxiety Inventory (BAI) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The BAI is a 21-item self-report measure used to rate subjective, somatic, and panic-related symptoms of anxiety on a scale of 0 to 3 (higher scores indicating more anxiety).
Change from Baseline in Anxiety Assessed by the Overall Anxiety Severity and Impairment Scale (OASIS) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The OASIS is a brief 5-item measure used to evaluate the functional impairment cause by anxiety; the frequency and intensity of anxiety, as well as the degree of avoidance and interference with work and social function are rated on a scale of 0 to 4 (higher scores indicating more anxiety).

SECONDARY OUTCOMES:
Change from Baseline in Pain Assessed by the Brief Pain Inventory (BPI) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The BPI contains 9 questions that assess the severity of pain, how much relief is provided by treatment, and the functional impact of the pain within the last 24 hours. Lower scores are better.
Change from Baseline in Pain Assessed by a Visual Analog Scale (VAS) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The VAS is a 100mm line where patients draw a vertical line to indicate their pain level from 0-100. Lower scores are better.
Change from Baseline in Pain Assessed by the Pain Distress Scale (PDS) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The PDS is an 11-point scale one where patients rate their pain by level of distress the pain causes on a scale of 0 to 10. Lower scores are better.
Change from Baseline in Pain Assessed by the Pain Disability Index (PDI) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  On the PDI, the patient rates how their pain affects 7 different areas of their life on a scale of the level of disability that their pain causes, from "no disability" to "worst disability". Lower scores are better.
Change from Baseline in Sleep Quality Assessed by the Pittsburgh Sleep Quality Index (PSQI) | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The PSQI contains 19 self-rated questions that assess sleep quality and disturbance over the previous 1-month period. The 19 items yield seven component scores such as sleep latency, sleep duration, and daytime dysfunction, which are then summed to generate a global score (higher scores indicating decreased sleep quality).
Change from Baseline in Quality of Life Assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The EORTC QLQ-C30 contains 30 questions assessing a cancer patient's quality of life. Lower scores indicate better quality of life and fewer symptoms.
Change from Baseline in Quality of Life Assessed by the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-BN20 | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The EORTC QLQ-BN20 module contains 20 additional questions specifically for brain tumor patients. Lower scores indicate better quality of life and fewer symptoms.
Patient's Global Impression of Change (PGIC) at Follow-Up | 1 week, 2 weeks, 4 weeks, 6 weeks, 8 weeks
  The PGIC is a single-question, 7-point scale depicting a patient's rating of overall improvement from "very much worse" to "very much improved".

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco Brain Tumor Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided